CLINICAL TRIAL: NCT01661634
Title: Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Ularitide (Urodilatin) Intravenous Infusion in Patients Suffering From Acute Decompensated Heart Failure [TRUE-AHF]
Brief Title: Efficacy and Safety of Ularitide for the Treatment of Acute Decompensated Heart Failure
Acronym: TRUE-AHF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cardiorentis (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ULA01; 2010-024249-59 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-09 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute decompensated heart failure
MeSH Terms: interventions — Ularitide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ularitide (Experimental): Ularitide, lyophilizate for i.v. infusion, 15 ng/kg BW/min, for 48 hours
  Interventions: Drug: Ularitide
- Placebo (Placebo Comparator): Placebo lyophilizate for i.v. infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ularitide
  Arms: Ularitide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a continuous intravenous (IV) ularitide infusion on the clinical status and outcome of patients with acute decompensated heart failure (ADHF).

DETAILED DESCRIPTION:
The objective of the TRUE-AHF study is to evaluate the effect of a 48-h continuous IV infusion of ularitide (15 ng/kg/min) versus placebo on the clinical status of patients with acute decompensated heart failure (ADHF).

The study drug will be administered in addition to the standard treatment. The nature of standard therapy will be carried out according to the clinical judgment of the Investigator and may include vasodilator, inotropic, and diuretic drugs, as clinically indicated.

There are two co-primary endpoints for this study. Co-primary endpoint 1 will be a hierarchical clinical composite variable that includes a patient-centered assessment of clinical progress, an assessment of lack of improvement or worsening of HF requiring a pre-specified intervention, and death.

The endpoint is intended to mimic the assessment that would be carried out by a physician caring for the patient. If, during the 48 h infusion, a patient's clinical course deteriorates because he/she dies, fails to improve or develops worsening HF requiring a pre-specified intervention or if the patient considers his/her general clinical status as moderately or markedly worse, the patient will be considered to be "worse". If the patient considers his/her general clinical status as moderately or markedly improved and if such improvement is sustained without fulfilling the criteria for "worse" throughout the 48-h infusion (from 0 h to 48 h), the patient will be considered to be "improved". If the patient is neither improved nor worse, the patient's clinical status will be considered to be "unchanged".

Co-primary efficacy endpoint 2 evaluates freedom from cardiovascular mortality during follow up after randomization, for the entire duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 85 years.
2. Unplanned hospitalization or emergency department visit for ADHF. Acute HF is defined as including all of the following:

   * Dyspnea at rest in a recumbent sitting position (30 to 45 degrees), which has worsened within the past week;
   * Radiological evidence of HF on a chest X-ray (if an appropriate chest;
   * computerized tomography scan is done; the X-ray need not be performed);
   * Brain natriuretic peptide (BNP) >500 pg/mL or NT-pro BNP >2000 pg/mL.
3. Ability to start infusion of the study drug within 12 h after initial clinical assessment.
4. Ability to reliably carry out self-assessment of symptoms.
5. Systolic blood pressure ≥116 mmHg and ≤180 mmHg at the time of randomization.
6. Persisting dyspnea at rest despite standard background therapy for ADHF (as determined by the Investigator) which must include IV furosemide (or equivalent diuretic) at ≥40 mg (or its equivalent) at any time after start of emergency services (ambulance, emergency department, or hospital). At the time of randomization, the patient must still be symptomatic. In addition, the patient should not have received an IV bolus of a diuretic for at least 2 h prior to randomization, and the infusion rates of all ongoing IV infusions of medications to treat HF must not have been increased or decreased for at least 2 h prior to randomization.
7. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local privacy regulations).

Exclusion Criteria:

1. Known active myocarditis, obstructive hypertrophic cardiomyopathy, congenital heart disease, restrictive cardiomyopathy, constrictive pericarditis, uncorrected clinically significant primary valvular disease.
2. Treatment with dobutamine at a dose >5 μg/kg/min or use of drugs for support of BP at the time of randomization.
3. Treatment with levosimendan, milrinone, or any other phosphodiesterase inhibitor within 7 days before randomization.
4. Treatment with nesiritide within 30 days before randomization.
5. Creatinine clearance <25 mL/min/1.73m² (as measured by the MDRD formula) at the time of screening.
6. Planned coronary revascularization procedure (percutaneous coronary intervention or coronary artery bypass grafting) within 5 days of randomization.
7. Clinical diagnosis of acute coronary syndrome meeting any 2 of the following 3 criteria:

   1. Prolonged chest pain at rest, or an accelerated pattern of angina
   2. Electrocardiogram changes indicative of ischemia or myocardial injury defined as: a new ST elevation at the J point of two anatomically contiguous leads with the cut-off points: ≥0.2 mV in men ≥40 years (>0.25 mV in men <40 years) or ≥0.15 mV in women in leads V2-V3 and/or ≥0.1 mV in other leads; or ST depression and T wave changes. New horizontal or down sloping ST depression ≥0.05 mV in two contiguous leads; and/or new T inversion ≥0.3 mV in two contiguous leads.
   3. Serum troponin >3 times upper limit of normal.
8. Clinically suspected acute mechanical cause of ADHF (e.g., papillary muscular rupture). The diagnosis need not be confirmed by imaging or cardiac catheterization.
9. Anemia (hemoglobin <9 g/dL or a hematocrit <25%).
10. Known vasculitis, active infective endocarditis, or suspected infections, e.g., pneumonia, acute hepatitis, systemic inflammatory response syndrome, or sepsis.
11. Body temperature ≥38°C just prior to randomization.
12. Acute or chronic respiratory disorder (e.g., severe chronic obstructive pulmonary disease) or primary pulmonary hypertension sufficient to cause dyspnea at rest, which may interfere with the ability to interpret dyspnea assessments or hemodynamic measurements.
13. Terminal illness other than congestive HF with expected survival <180 days.
14. Any previous exposure to ularitide.
15. Known allergy to natriuretic peptides.
16. Participation in an investigational clinical drug study within 30 days prior to randomization.
17. Current drug abuse or chronic alcoholism sufficient to impair participation and compliance to the study protocol.
18. Women who are breast-feeding.
19. Women of child-bearing potential (i.e., pre-menopausal women) without documentation of a negative urine/blood pregnancy assay within 12 h prior to randomization.
20. Any condition that, in the Investigator's opinion, makes the patient unsuitable for study participation.
21. Legal incapacity or limited legal capacity.
22. Patients requiring mechanical circulatory support.
23. Patients with severe hepatic impairment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2157 (Actual)
Dates: Start 2012-07; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Two Co-primary Efficacy Endpoints | 6, 24, 48 hours post infusion through the entire duration of the trial
  Improvement in a hierarchical clinical composite comprised of elements associated with: patient global assessment using a 7-point scale of symptomatic improvement, lack of improvement, or worsening; persistent or worsening heart failure (HF) requiring an intervention (initiation or intensification of IV therapy, circulatory or ventilatory mechanical support, surgical intervention, ultrafiltration, hemofiltration or dialysis); and all-cause mortality. Assessment of the clinical composite will be performed at 6 hour (h), 24 h and 48 h after start of IV ularitide infusion
  Freedom from cardiovascular mortality during follow up after randomization, for the entire duration of the trial.

SECONDARY OUTCOMES:
Length of stay of index hospitalization in hours after start of study drug infusion | up to 30 days
Length of stay in intensive care (intensive care unit [ICU] or critical care unit [CCU]) | during the first 120 h following the start of the study drug infusion.
Number of events of persistent or worsening HF requiring an intervention | from the start of the study drug infusion to 120 h.
Proportion of patients with persistent or worsening HF and requiring an intervention | from the start of study drug infusion to 120 h.
Reduction in rehospitalization for heart failure | within 30 days after initial hospital
Changes of N-terminal pro brain natriuretic peptide (NT-pro BNP) | 48 h of treatment compared to baseline.
Time to completion of last dose of any IV drugs that can be used for the treatment of HF (e.g., diuretics, vasodilators, or positive inotropic agents) | for the first 120 h following the start of the drug infusion.
Change in serum creatinine | from baseline through 72 h.
180 days after start of study drug infusion, including patients still hospitalized at Day 30. | All-cause mortality and cardiovascular rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Milton Packer, MD, Study Chair; Christopher O'Connor, MD, Principal Investigator; William F. Peacock, MD, Principal Investigator
Locations (138):
- United States (37):
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Sacramento, California
  - Littleton, Colorado
  - Trumbull, Connecticut
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Lawrenceville, Georgia
  - Peoria, Illinois
  - Rockford, Illinois
  - Kansas City, Kansas
  - Alexandria, Louisiana
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Newark, New Jersey
  - Brooklyn, New York
  - The Bronx, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Middletown, Ohio
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Norfolk, Virginia
  - Salem, Virginia
- Argentina (11):
  - Ciudad Autonoma, Buenos Aires
  - Coronel Suárez, Buenos Aires
  - La Plata, Buenos Aires
  - Córdoba, Córdoba Province
  - San Vicente, Córdoba Province
  - Rosario, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Corrientes
  - Córdoba
  - San Miguel de Tucumán
  - Santa Fe
- Belgium (2):
  - Aalst
  - Kortrijk
- Brazil (5):
  - Goiânia, Goiás
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
- Canada (2):
  - Halifax, Nova Scotia
  - Montreal, Quebec
- Czechia (6):
  - Brno
  - Frýdek-Místek
  - Hradec Králové
  - Olomouc
  - Prague
  - Znojmo
- Tallinn, Estonia
- Espoo, Finland
- France (6):
  - Besançon, Doubs
  - Toulouse, Haute Garonne
  - Paris, Paris
  - Bayonne, Pyrenees Atlantiques
  - Bron, Rhone
  - Poitiers, Vienne
- Germany (9):
  - Nuremberg, Bavaria
  - Bad Nauheim, Hesse
  - Groß-Umstadt, Hesse
  - Langen, Hesse
  - Greifswald, Mecklenburg-Vorpommern
  - Bochum, North Rhine-Westphalia
  - Erfurt, Thuringia
  - Jena, Thuringia
  - Berlin
- Debrecen, Hungary
- Israel (8):
  - Afula
  - Ashkelon
  - Hadera
  - Holon
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Safed
- Italy (13):
  - San Fermo della Battaglia, Como
  - Legnano, Milano
  - Rozzano, Milano
  - Alessandria
  - Bari
  - Bologna
  - Como
  - Genova
  - Milan
  - Napoli
  - Novara
  - Roma
  - Varese
- Riga, Latvia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Netherlands (6):
  - Beverwijk
  - Ede
  - Gorinchem
  - Groningen
  - Leiderdorp
  - Sneek
- Poland (4):
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
- Romania (3):
  - Bucharest
  - Iași
  - Oradea
- Serbia (5):
  - Belgrade
  - Kamenitz
  - Niš
  - Niška Banja
  - Zemun
- Spain (8):
  - L'Hospitalet de Llobregat, Barcelona
  - Sant Joan Despí, Barcelona
  - Santiago de Compostela, La Coruña
  - Aranjuez, Madrid
  - Majadahonda, Madrid
  - Alicante
  - Barcelona
  - Madrid
- Switzerland (3):
  - Basel
  - Lugano
  - Zurich
- Turkey (Türkiye) (4):
  - Eskişehir
  - Istanbul
  - Kocaeli
  - Sivas

REFERENCES:
- [Background] Mitrovic V, Luss H, Nitsche K, Forssmann K, Maronde E, Fricke K, Forssmann WG, Meyer M. Effects of the renal natriuretic peptide urodilatin (ularitide) in patients with decompensated chronic heart failure: a double-blind, placebo-controlled, ascending-dose trial. Am Heart J. 2005 Dec;150(6):1239. doi: 10.1016/j.ahj.2005.01.022. PMID 16338265
- [Background] Mitrovic V, Seferovic PM, Simeunovic D, Ristic AD, Miric M, Moiseyev VS, Kobalava Z, Nitsche K, Forssmann WG, Luss H, Meyer M. Haemodynamic and clinical effects of ularitide in decompensated heart failure. Eur Heart J. 2006 Dec;27(23):2823-32. doi: 10.1093/eurheartj/ehl337. Epub 2006 Oct 30. PMID 17074775
- [Derived] Packer M, O'Connor C, McMurray JJV, Wittes J, Abraham WT, Anker SD, Dickstein K, Filippatos G, Holcomb R, Krum H, Maggioni AP, Mebazaa A, Peacock WF, Petrie MC, Ponikowski P, Ruschitzka F, van Veldhuisen DJ, Kowarski LS, Schactman M, Holzmeister J; TRUE-AHF Investigators. Effect of Ularitide on Cardiovascular Mortality in Acute Heart Failure. N Engl J Med. 2017 May 18;376(20):1956-1964. doi: 10.1056/NEJMoa1601895. Epub 2017 Apr 12. PMID 28402745
- [Derived] Packer M, Holcomb R, Abraham WT, Anker S, Dickstein K, Filippatos G, Krum H, Maggioni AP, McMurray JJV, Mebazaa A, O'Connor C, Peacock F, Ponikowski P, Ruschitzka F, van Veldhuisen DJ, Holzmeister J; TRUE-AHF Investigators and Committees. Rationale for and design of the TRUE-AHF trial: the effects of ularitide on the short-term clinical course and long-term mortality of patients with acute heart failure. Eur J Heart Fail. 2017 May;19(5):673-681. doi: 10.1002/ejhf.698. Epub 2016 Nov 13. PMID 27862700